CLINICAL TRIAL: NCT04133415
Title: A Trial of Palliative Lattice Stereotactic Body Radiotherapy (SBRT)
Brief Title: Palliative Lattice Stereotactic Body Radiotherapy (SBRT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201910071
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Cancer; Palliative Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lattice stereotactic body radiation therapy (Experimental): -Lattice SBRT prescribed to a dose of 20 Gy in 5 fractions with a simultaneous integrated boosts of 66.7 Gy in 5 fractions
  Interventions: Radiation: Lattice stereotactic body radiation therapy; Procedure: Peripheral blood

INTERVENTIONS:
Radiation: Lattice stereotactic body radiation therapy — -As long as radiotherapy fields do not overlap, treatment of up to 4 other tumor sites are allowed
  Other Names: Lattice SBRT
Procedure: Peripheral blood — -Before treatment, immediately after radiotherapy completion, 14 days after radiotherapy, and 30 days after radiotherapy

SUMMARY:
Standard palliative radiotherapy regimens may provide limited durability of response in large tumors. Thus, there is a clinical need for a new approach. The Lattice SBRT approach will deliver 20 Gy in 5 fractions with partial volume simultaneous integrated boosts to 66.7 Gy. This is hypothesized to improve symptom response, local control, and better prime the tumor microenvironment for immune response compared with standard palliative radiotherapy doses. It is also hypothesized that this will be associated with less toxicity than the traditional homogenous SBRT plan delivered to a large tumor. Blood will be collected before and after Lattice SBRT for evaluation of the peripheral blood immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cancer.
* Planning to undergo palliative radiotherapy to a lesion ≥ 4.5 cm as measured with radiographic imaging or with calipers by clinical exam.
* ECOG performance status ≤ 2
* At least 18 years of age.
* Radiotherapy is known to be teratogenic. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior radiotherapy that overlaps with any planned site of protocol radiotherapy.
* Patients with tumors in need of urgent surgical intervention, such as life-threatening bleeding or those at high risk for pathologic fracture.
* Currently receiving any cytotoxic cancer therapy regimens or VEGF inhibitors that will overlap with the Lattice SBRT administration.

  *Cytotoxic chemotherapy and VEGF inhibitors prior to radiotherapy or planned after radiotherapy delivery are allowed at the discretion of the treating radiation oncologist. This includes continuing a treatment plan which was initiated prior to the start of radiotherapy. A 2 week washout is recommended, but not required.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 20 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spraker, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duriseti S, Kavanaugh J, Goddu S, Price A, Knutson N, Reynoso F, Michalski J, Mutic S, Robinson C, Spraker MB. Spatially fractionated stereotactic body radiation therapy (Lattice) for large tumors. Adv Radiat Oncol. 2021 Jan 8;6(3):100639. doi: 10.1016/j.adro.2020.100639. eCollection 2021 May-Jun. PMID 34195486
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lattice Stereotactic Body Radiation Therapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lattice Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 64 [30 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Treatment-related, Non-hematologic, Grade 3 or Higher Adverse Events
Description: -Measured by CTCAE version 5.0
Time Frame: Through 90 days following completion of radiotherapy (estimated to be 90 days and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Lattice Stereotactic Body Radiation Therapy
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 90 days following completion of treatment.
Arm/Group | Lattice Stereotactic Body Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 6/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lattice Stereotactic Body Radiation Therapy (N=20)
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lattice Stereotactic Body Radiation Therapy (N=20)
Anemia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
COVID-19 (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dypsnea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT04133415/Prot_SAP_000.pdf